CLINICAL TRIAL: NCT05765370
Title: LDL Cholesterol TARGETs in OLDer Patients (Age≥75 Years) With Atherosclerotic Cardiovascular Disease (TARGET OLD)
Brief Title: LDL Cholesterol TARGETs in OLDer Patients (Age≥75 Years) With ASCVD (TARGET OLD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-1879
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Atherosclerotic Cardiovascular Disease; Older Patients; LDL Cholesterol
Keywords: LDL-C target; Atherosclerotic Cardiovascular Disease; Older patients; Age≥75 years; Lipid-lowering therapy; Stain; PCSK9 inhibitor
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants and study investigators were aware of the study-group assignments, but outcome adjudicators were not. All potential cardiovascular events and safety events were adjudicated according to prespecified criteria by an independent clinical events committee whose members were unaware of the trial-group assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LDL-C Lower-Target Group (25mg/dL≤ LDL-C<70mg/dL) (Experimental): Participants randomized into the LDL-C lower-target arm will have a goal of 25mg/dL≤ LDL-C<70mg/dL.
  Prescription of lipid-lowering agents (drug and dosage) were initiated or adjusted on the basis of the investigator according to the assigned target LDL-C level.
  Interventions: Procedure: Achieving a Target LDL-C level of 25mg/dL≤ LDL-C<70mg/dL
- LDL-C Higher-Target Group (70mg/dL≤ LDL-C<100mg/dL) (Active Comparator): Participants randomized into the LDL-C lower-target arm will have a goal of 70mg/dL≤ LDL-C<100mg/dL.
  Prescription of lipid-lowering agents (drug and dosage) were initiated or adjusted on the basis of the investigator according to the assigned target LDL-C level.
  Interventions: Procedure: Achieving a Target LDL-C level of 70mg/dL≤ LDL-C<100mg/dL

INTERVENTIONS:
Procedure: Achieving a Target LDL-C level of 25mg/dL≤ LDL-C<70mg/dL — Investigators initiated or adjusted lipid-lowering agents (drug and dosage) to achieve the target of 25mg/dL≤ LDL-C<70mg/dL. The protocol encouraged, but did not mandate, the initiation of moderate-intensity statin therapy for secondary prevention with the evaluation of the potential for ASCVD risk reduction, adverse effects, and drug-drug interactions, as well as patient frailty and patient preferences. Statin monotherapy or in combination with ezetimibe, PCSK9 inhibitor or other drugs were adjusted on the basis of LDL-C levels.
  At each follow-up visit, the investigators should verify whether the target LDL-C has been obtained. If the target level of LDL cholesterol was achieved, it is reasonable to continue to monitor adherence to lifestyle modiﬁcations, medication, and ongoing LDL-C response to therapy. If the target level of LDL cholesterol was not achieved, adjustment of the type and dose regimen of statin, or the additional of a nonstatin agent should be considered.
  Arms: LDL-C Lower-Target Group (25mg/dL≤ LDL-C<70mg/dL)
Procedure: Achieving a Target LDL-C level of 70mg/dL≤ LDL-C<100mg/dL — Investigators initiated or adjusted lipid-lowering agents (drug and dosage) to achieve the target of 70mg/dL≤ LDL-C<100mg/dL. The protocol encouraged, but did not mandate, the initiation of moderate-intensity statin therapy for secondary prevention with the evaluation of the potential for ASCVD risk reduction, adverse effects, and drug-drug interactions, as well as patient frailty and patient preferences. Statin monotherapy or in combination with ezetimibe, PCSK9 inhibitor or other drugs were adjusted on the basis of LDL-C levels.
  At each follow-up visit, the investigators should verify whether the target LDL-C has been obtained. If the target level of LDL cholesterol was achieved, it is reasonable to continue to monitor adherence to lifestyle modiﬁcations, medication, and ongoing LDL-C response to therapy. If the target level of LDL cholesterol was not achieved, adjustment of the type and dose regimen of statin, or the additional of a nonstatin agent should be considered.
  Arms: LDL-C Higher-Target Group (70mg/dL≤ LDL-C<100mg/dL)

SUMMARY:
To determine whether treating to an LDL-C target of 25 to <70 mg/dL is superior to an LDL-C target of 70 to <100 mg/dL with respect to major cardiovascular events (cardiovascular death, myocardial infarction, stroke, hospitalization for unstable angina, or coronary revascularization) in patients aged ≥75 years with atherosclerotic cardiovascular disease (ASCVD).

To determine whether treating to an LDL-C target of 25 to <70 mg/dL is non-inferior to an LDL-C target of 70 to <100 mg/dL with respect to major safety events (hemorrhagic stroke, new-onset diabetes, muscle-related events, neurocognitive adverse events, new or recurrent cancer, cataract, or hepatic disorder [Alanine aminotransferase (ALT)/Aspartate aminotransferase (AST) >3× ULN, or total bilirubin >2× ULN]) in patients aged ≥75 years with ASCVD.

DETAILED DESCRIPTION:
The benefits of LDL cholesterol-lowering treatment for the prevention of atherosclerotic cardiovascular disease (ASCVD) are well established. LDL-C lowering is associated with a significant reduction in major adverse cardiovascular events in a linear fashion, apparently without any plateau at low LDL-C levels. On the other hand, the degree to which LDL-C levels can be safely lowered remains unclear. It is still controversial whether lower LDL-C levels are associated with signiﬁcant clinical adverse effects (e.g. new-onset diabetes mellitus or possibly hemorrhagic stroke) and long-term data are needed to address safety concerns.

It should be noted that the benefits and risks from LDL cholesterol lowering in older patients (age ≥75 years) remains debated because most randomized trials have explicitly excluded or enrolled few older adults. In clinical practice, the appropriate treatment target for LDL-C in patients ≥75 years of age with ASCVD remains uncertain. Current US and European cholesterol guidelines have no specific recommendations regarding the LDL-C treatment goal for older patients and noted that the level of evidence in older patients is low. Currently, there is no direct evidence from randomized clinical trials (RCTs) for the most appropriate treatment targets for LDL-C among patients ≥75 years of age with ASCVD in worldwide.

The TARGET OLD trial is a multicenter, open-label, parallel-group, event-driven, randomized, controlled trial with blinded end-point evaluation. Consecutive patients aged ≥75 years with ASCVD who meet the inclusion criteria and none of the exclusion criteria outlined above will be randomized in a 1:1 fashion to LDL-C target of 25 to <70 mg/dL or LDL-C target of 70 to <100 mg/dL. The proposed study will examine the comparative efficacy and safety of treating to an LDL-C target of 25 to <70 mg/dL compared with an LDL-C target of 70 to <100 mg/dL among patients aged 75 years or older with ASCVD. Our primary hypothesis is that, among such patients, targeting an LDL-C of 25 to less than 70 mg/dL is superior to a target of 70 to less than 100 mg/dL on reducing the risk of major adverse cardiovascular events (primary efficacy end point), while is non-inferior towards the composite of major safety outcomes (key secondary safety end point).

Prescription of lipid-lowering agents (drug and dosage up to the investigator according to the assigned target LDL-C level. Statin monotherapy or in combination with ezetimibe, PCSK9 inhibitor or other drugs were adjusted on the basis of the study-group assignment. Patients will follow-up at 1, 2, 4, 6, 12 months, and then every 6 months throughout 36 months with an evaluation of patients' lipid profiles, any cardiovascular events, safety and adverse events, muscle-related symptoms, quality of life (EQ-5D), and patient-reported cognition function (ECog scale). The trial will continue until 726 adjudicated primary endpoint events have occurred. We estimated that 4,200 patients would be needed to provide the necessary number of confirmed endpoints to test the study hypothesis. All analyses will be according to the intention-to-treat (ITT) principle.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥75 years of age
2. Diagnosis of clinical atherosclerotic cardiovascular disease (ASCVD) with one or more of the following:

   1. Diagnosis of coronary heart disease (one or more of the following criteria must be satisfied):

      * Hospitalization for acute coronary syndrome
      * Treatment or hospitalization for stable angina pectoris with documented ischemia on invasive or noninvasive testing
      * History of myocardial infarction
      * History of coronary revascularization procedure (eg, percutaneous coronary intervention [PCI] or coronary artery bypass graft surgery [CABG])
      * Invasive diagnostic coronary angiography indicating >50% stenosis in at least one major epicardial coronary artery or CT-imaging (eg, CCTA/MDCT) evidence of coronary atherosclerosis (>50% stenosis in at least two major epicardial coronary artery)
   2. Diagnosis of atherosclerotic cerebrovascular or carotid disease (one or more of the following criteria must be satisfied):

      * History of ischemic stroke or transient ischemic attack (TIA) confirmed by symptoms with a documented ischemic lesion on CT or MRI in the cerebral regions corresponding to the symptoms;
      * Documented intracranial atherosclerotic stenosis on the basis of conventional cerebral angiography, magnetic resonance angiography, CT angiography, transcranial doppler ultrasound, and high-resolution MRI;
      * Symptomatic carotid artery disease with ≥50% carotid arterial stenosis;
      * Asymptomatic carotid artery disease with ≥70% carotid arterial stenosis per angiography or duplex ultrasound;
      * History of carotid revascularization (catheter-based or surgical).
   3. Diagnosis of atherosclerotic peripheral artery disease (one or more of the following criteria must be satisfied):

      * History of aorto-iliac or peripheral arterial intervention (catheter-based or surgical).
      * Prior non-traumatic amputation of a lower extremity due to peripheral artery disease
      * History of intermittent claudication and one or more of the following:

        1. An ankle/arm blood pressure (BP) ratio < 0.90, or
        2. Significant peripheral artery stenosis (≥50%) documented by angiography, or by duplex ultrasound
3. Baseline LDL-C level should be satisfied:

   * Patients were required to have a baseline LDL-C level ≥100mg/dL (2.6mmol/L) if they were taking a regimen of lipid-lowering therapy <4 weeks or they had not previously received lipid-lowering therapy.
   * Patients were required to have a baseline LDL-C level ≥70mg/dL (1.8mmol/L) if they were on stable treatment with lipid-lowering therapy ≥4 weeks
4. Signed written informed consent.

Exclusion Criteria:

1. Subject was clinically unstable:

   1. Hypotension, defined as sustained systolic blood pressure of <90 mmHg due to cardiac failure with associated symptoms;
   2. Unstable or severe pulmonary edema/decompensated congestive heart failure;
   3. Acute mitral regurgitation or acute ventricular septal defect;
   4. Cardiogenic shock and/or need for mechanical/pharmacologic hemodynamic support
   5. Ongoing Non-STEMI with biomarkers (cardiac troponin) still rising
   6. Recent STEMI (≤7 days prior to randomization)
   7. Recurrent symptoms of cardiac ischemia
2. Moderate to severe heart failure (New York Heart Association [NYHA] Functional Classiﬁcation III or IV) or last known left ventricular ejection farction (LVEF) <40%.
3. Severe renal dysfunction, deﬁned as creatinine clearance <30 mL/min or estimated glomerular filtration (eGFR) rate less than 30 ml/min/1.73 m2, or requirement for peritoneal dialysis or hemodialysis for renal insufficiency.
4. History of hemorrhagic stroke or unknown classified stroke.
5. Uncontrolled or recurrent ventricular tachycardia (such as ventricular fibrillation, recurrent and highly symptomatic ventricular tachycardia, complete heart block, atrial ﬁbrillation with rapid ventricular response, or supraventricular tachycardia that are not controlled by medications).
6. Uncontrolled hypertension (greater than 180 mm Hg systolic and/or greater than 110 mm Hg diastolic at randomization visit).
7. History or clinical evidence of active liver disease or hepatic dysfunction, deﬁned as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 × upper limit of normal (ULN), or total bilirubin > 2 × ULN.
8. Unexplained elevated creatine kinase (CK) concentration >5 × ULN or elevation due to known muscle disease.
9. Planned or expected cardiac surgery, PCI or carotid stenting, or planned major noncardiac surgery during the study period. If angiography or revascularization is planned, patients may be screened and enrolled after all such planned procedures are completed.
10. Active Malignancy (except nonmelanoma skin cancers, cervical in-situ carcinoma, breast ductal carcinoma in situ, or stage 1 prostate carcinoma) including those patients requiring surgery, chemotherapy, and/or radiation in the past 3 years.
11. Drug or alcohol abuse, and inability/unwillingness to abstain from drug abuse and excessive alcohol consumption during the study.
12. Severe, concomitant noncardiovascular disease that is expected to reduce life expectancy to <3 years
13. Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(ies), or receiving other investigational agent(s)
14. Subject has received drugs via a systemic route that have known major interactions with background statin therapy (eg, itraconazole, ketoconazole, and other antifungal azoles, erythromycin, clarithromycin, or cyclosporine nefazodone) within 1 month prior to randomization or is likely to require such treatment during the study period.
15. Recipient of any major organ transplant (eg, lung, liver, heart, bone marrow, renal)
16. Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (eg, Clinical Outcome Assessments) to the best of the subject and investigator's knowledge.
17. Any uncontrolled or serious disease, or any medical or surgical condition (such as known active infection or major hematologic, renal, metabolic, gastrointestinal or endocrine dysfunction, or a chronic disease or infection [eg, HIV]), that may either interfere with participation in the clinical study and is not currently stable and appropriately managed in the judgment of the investigator, and/or put the subject at significant risk (according to investigator's judgment) if he/she participates in the clinical study.
18. Mental/psychological impairment/neurocognitive disorder, or any other reason to expect patient difficulty in complying with the requirements of the study or understanding the goal and potential risks of participating in the study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4200 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2026-09-24 (Estimated); Study Completion 2026-12-24 (Estimated)

PRIMARY OUTCOMES:
Time to first occurrence of major cardiovascular events (composite of cardiovascular death, myocardial infarction, stroke, hospitalization for unstable angina, coronary revascularization) | From randomization until study completion (until 726 adjudicated primary endpoint events have occurred); for approximately a median follow-up of 42 months
  The primary endpoint measure was the number of patients with a first occurrence of adjudicated composite of cardiovascular death, myocardial infarction, stroke, hospitalization for unstable angina, or coronary revascularization during the follow-up period.

SECONDARY OUTCOMES:
Time to first occurrence of major safety events (composite of hemorrhagic stroke, new-onset diabetes, muscle-related events, neurocognitive adverse events, new or progressive cancer, cataract, or hepatic disorder). | From randomization until study completion (until 726 adjudicated primary endpoint events have occurred); for approximately a median follow-up of 42 months
  The key secondary endpoint measure was the number of patients with a first occurrence of adjudicated composite of hemorrhagic stroke, new-onset diabetes, muscle-related events, neurocognitive adverse events, new or progressive cancer, cataract, or hepatic disorder (ALT/AST >3× ULN, or total bilirubin >2× ULN) during the follow-up period.
Time to first occurrence of composite endpoint of cardiovascular death, myocardial infarction, stroke, or coronary revascularization. | From randomization until study completion (until 726 adjudicated primary endpoint events have occurred); for approximately a median follow-up of 42 months.
  Number of patients with a first occurrence of adjudicated composite of cardiovascular death, myocardial infarction, stroke, or coronary revascularization during the follow-up period.
Time to first occurrence of composite endpoint of cardiovascular death, myocardial infarction, or stroke. | From randomization until study completion (until 726 adjudicated primary endpoint events have occurred); for approximately a median follow-up of 42 months.
  Number of patients with a first occurrence of adjudicated composite of cardiovascular death, myocardial infarction, or stroke during the follow-up period.
Time to first occurrence of composite endpoint of all-cause death, myocardial infarction, or stroke. | From randomization until study completion (until 726 adjudicated primary endpoint events have occurred); for approximately a median follow-up of 42 months.
  Number of patients with a first occurrence of adjudicated composite of all-cause death, myocardial infarction, or stroke during the follow-up period.
Time to first occurrence of composite endpoint of cardiovascular death or myocardial infarction. | From randomization until study completion (until 726 adjudicated primary endpoint events have occurred); for approximately a median follow-up of 42 months.
  Number of patients with a first occurrence of adjudicated composite of cardiovascular death or myocardial infarction during the follow-up period.
Time to first occurrence of composite endpoint of all-cause death or myocardial infarction. | From randomization until study completion (until 726 adjudicated primary endpoint events have occurred); for approximately a median follow-up of 42 months.
  Number of patients with a first occurrence of adjudicated composite of all-cause death or myocardial infarction during the follow-up period.
Time to first occurrence of myocardial infarction. | From randomization until study completion (until 726 adjudicated primary endpoint events have occurred); for approximately a median follow-up of 42 months.
  Number of patients with a first occurrence of adjudicated myocardial infarction during the follow-up period.
Time to first occurrence of coronary revascularization. | From randomization until study completion (until 726 adjudicated primary endpoint events have occurred); for approximately a median follow-up of 42 months.
  Number of patients with a first occurrence of adjudicated coronary revascularization during the follow-up period.
Time to cardiovascular death. | From randomization until study completion (until 726 adjudicated primary endpoint events have occurred); for approximately a median follow-up of 42 months.
  Number of patients with an occurrence of cardiovascular death during the follow-up period.
Time to first occurrence of stroke. | From randomization until study completion (until 726 adjudicated primary endpoint events have occurred); for approximately a median follow-up of 42 months.
  Number of patients with a first occurrence of stroke during the follow-up period.
Time to first occurrence of hospitalization for unstable angina. | From randomization until study completion (until 726 adjudicated primary endpoint events have occurred); for approximately a median follow-up of 42 months.
  Number of patients with a first occurrence of hospitalization for unstable angina during the follow-up period.
Time to all-cause death. | From randomization until study completion (until 726 adjudicated primary endpoint events have occurred); for approximately a median follow-up of 42 months.
  Number of patients with an occurrence of all-cause death during the follow-up period.

OTHER OUTCOMES:
Health-related Quality-of-life outcome | Baseline, 30 days, 6 months, 1 year, and then every 6 months until study completion (726 adjudicated primary endpoint events have occurred)
  Quality of life as measured by European Quality of Life-5 Dimensions (EQ-5D-5L)
Patient-reported cognition function | Baseline, 30 days, 6 months, 1 year, and then every 6 months until study completion (726 adjudicated primary endpoint events have occurred).
  Patient-reported cognition function as measured by Everyday Cognition (ECog) scale

CONTACTS AND LOCATIONS:
Overall Officials: Kefei Dou, MD, PhD, Principal Investigator — Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing; Hao-Yu Wang, MD, PhD, Principal Investigator — Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No